CLINICAL TRIAL: NCT03771066
Title: Randomized Trial Examining Oral Consumption of Bisphenol A on Type 2 Diabetes Risk Markers
Brief Title: Bisphenol A and Muscle Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Todd Hagobian, Associate Professor, California Polytechnic State University-San Luis Obispo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-149-CP
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Insulin Sensitivity; Glucose Metabolism Disorders; Microtia
Keywords: bisphenol A; diet
MeSH Terms: conditions — Insulin Resistance; Glucose Metabolism Disorders; Congenital Microtia | interventions — bisphenol A

STUDY DESIGN:
Intervention Model Description: This experimental study is a 2-group randomized, clinical trial comparing a 4-day energy balance diet plus oral BPA consumption at 50 ug/kg body weight (Diet+BPA) vs. 4-day energy balance diet plus oral placebo consumption (Diet+No BPA). Forty participants will be randomized to Diet+BPA and Diet+No BPA and will reside in a supervised environment at Cal Poly's sleep research facilities for 6 days (2-day baseline run-in, followed by 4-day treatment). Main outcome measures (muscle insulin sensitivity and hepatic glucose suppression) will be assessed at baseline and treatment periods.
Who Masked: Participant, Outcomes Assessor
Masking Description: This study will be a double-blinded study. Research staff collecting data and participants will not know treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet plus bisphenol A (Experimental): Participants will receive a 4-day diet plus bisphenol A at 50 ug/kg body weight.
  Interventions: Behavioral: bisphenol A
- Placebo (Placebo Comparator): Participants will receive a 4-day diet plus no bisphenol A.
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: bisphenol A — Vanilla wafer cookie with bisphenol A administered
  Arms: Diet plus bisphenol A
Behavioral: Placebo — Vanilla wafer cookie with no bisphenol A
  Arms: Placebo

SUMMARY:
This study examine oral bisphenol A consumption on muscle insulin sensitivity and hepatic glucose suppression. Half of the participants will receive a diet plus BPA and the other half will receive a diet plus no bisphenol A.

DETAILED DESCRIPTION:
Evidence linking bisphenol A exposure with diabetes risk remains mainly associative in nature, and mechanism linking bisphenol A to type 2 diabetes remains unclear. The investigator's preliminary data suggests that in young adults, single oral BPA consumption significantly decreased glucose, insulin, and C-Peptide responses to an oral glucose tolerance test, suggesting that immediate consumption of bisphenol A has an effect on muscle insulin sensitivity, hepatic glucose suppression and/or digestion and absorption to lower blood glucose, insulin, and C-Peptide concentrations. The present experimental study evaluating the effects of bisphenol A over several days on the pathogenesis of type 2 diabetes will directly assess each of these potential mechanisms using gold standard measures (euglycemic hyperinsulinemic clamp technique and hepatic glucose suppression with glucose stable isotope infusion, and fecal microbiota).

ELIGIBILITY:
Inclusion Criteria:

* non-dieting
* sedentary (≤3 hour/week of aerobic exercise)
* normal-weight (BMI = 18.5 to 24.9 kg/m2)
* weight-stable for the previous 6 months
* free of any metabolic or chronic disease
* non-smoking, and sedentary

Exclusion Criteria:

* Hemoglobin A1C based on the American Diabetes Association guidelines of 5.7 to 6.4% (Prediabetes) or >6.4% (Diabetes)
* impaired glucose tolerance
* type 1 diabetes
* type 2 diabetes
* colitis or any inflammatory bowel condition
* neurologic or psychiatric conditions
* smoking
* special diets (e.g. vegetarian, low-carbohydrate, Paleolithic, etc.)
* pregnant women or women trying to become pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in rate of glucose disposal | Baseline and 4 days
  Three hour euglycemic hyperinsulinemic clamp technique with stable glucose isotope infusion to determine rate of glucose disposal
Change in rate of glucose appearance | Baseline and 4 days
  Ninety minutes stable glucose isotope infusion to determine rate of hepatic glucose appearance

SECONDARY OUTCOMES:
Change in concentration of insulin | Baseline and 4 days
  Fasting blood sample for insulin concentration
Change in concentration of glucose | Baseline and 4 days
  Fasting blood sample for glucose concentration
Change in concentration of c-peptide | Baseline and 4 days
  Fasting blood sample for c-peptide concentration
Change in concentration of proinsulin | Baseline and 4 days
  Fasting blood sample for proinsulin
Change in concentration of adiponectin | Baseline and 4 days
  Fasting blood sample for adiponectin
Change in concentration of 17-beta estradiol | Baseline and 4 days
  Fasting blood sample for 17-beta estradiol
Change in concentration of firmicutes | Baseline and 4 days
  Fecal microbiome concentration of firmicutes
Change in concentration of clostridia | Baseline and 4 days
  Fecal microbiome concentration of clostridia

CONTACTS AND LOCATIONS:
Overall Officials: Todd Hagobian, PhD, Principal Investigator — California Polytechnic State University-San Luis Obispo; Hannah Brunner-Gaydos, Study Director — California Polytechnic State University-San Luis Obispo
Locations (1):
- California Polytechnic State University, San Luis Obispo, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion, and will be available indefinitely.
Access Criteria: Data access will be freely available for download on the Cal Poly Digital Commons website. Requestors will be required to sign a data access agreement.
URL: https://digitalcommons.calpoly.edu

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT03771066/Prot_SAP_ICF_003.pdf